CLINICAL TRIAL: NCT06158945
Title: The Role of Endothelin 1 as a Marker of Renal Impairment in Sickle Cell Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Anwar Qenawy, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: soh_Med_23_10_01MS
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: urinary endothelin 1 — assesment of endothelin 1 in urinary sample

SUMMARY:
Sickle cell disease (SCD) refers to a group of hemoglobinopathies that include mutations in the gene encoding the beta subunit of hemoglobin. Within the umbrella of SCD, many subgroups exist, namely sickle cell anemia (SCA), hemoglobin SC disease (HbSC), and hemoglobin sickle-beta-thalassemia (beta-thalassemia positive or beta-thalassemia negative). Several other minor variants within the group of SCDs also, albeit not as common as the varieties mentioned above. It is essential to mention the sickle cell trait (HbAS), which carries a heterozygous mutation and seldom presents clinical signs or symptoms. Sickle cell anemia is the most common form of SCD

ELIGIBILITY:
Inclusion Criteria:

* The patients fulfilling all the following criteria will be included:
* Patients with sickle cell disease in the age range of 1-18years.

Exclusion Criteria:

* Patients diagnosed to have coexistent renal disease before the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patients fulfilling all the following criteria will be included:
  Patients with sickle cell disease in the age range of 1-18years
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-10-23 (Estimated); Study Completion 2024-10-23 (Estimated)

PRIMARY OUTCOMES:
renal affection in sickle cell patients | 1 year
  assessment of urinary endothelin 1 as a marker of renal impairment in sickle cell patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams TN, Thein SL. Sickle Cell Anemia and Its Phenotypes. Annu Rev Genomics Hum Genet. 2018 Aug 31;19:113-147. doi: 10.1146/annurev-genom-083117-021320. Epub 2018 Apr 11. PMID 29641911
- [Background] Platt OS. Sickle cell anemia as an inflammatory disease. J Clin Invest. 2000 Aug;106(3):337-8. doi: 10.1172/JCI10726. No abstract available. PMID 10930436
- [Background] Lonergan GJ, Cline DB, Abbondanzo SL. Sickle cell anemia. Radiographics. 2001 Jul-Aug;21(4):971-94. doi: 10.1148/radiographics.21.4.g01jl23971. PMID 11452073
- [Background] Nath KA, Katusic ZS. Vasculature and kidney complications in sickle cell disease. J Am Soc Nephrol. 2012 May;23(5):781-4. doi: 10.1681/ASN.2011101019. Epub 2012 Mar 22. PMID 22440903